CLINICAL TRIAL: NCT00201877
Title: A Phase II Study of Velcade (Bortezomib, PS-341) and Rituximab in Relapsed/Refractory Mantle Cell and Follicular Non-Hodgkin's Lymphoma
Brief Title: Velcade (Bortezomib, PS-341) and Rituximab in Relapsed/Refractory Mantle Cell and Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0430; NCI-2011-03233 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
Keywords: Relapsed/Refractory; NHL; Follicular; Mantle Cell; non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Recurrence | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade and Rituximab (Experimental): Rituximab 375 mg/m2 IV day 1 of weeks 4, 5, 7, 8, 10, 11, 13, and 14 prior to Velcade™ administration.
  Velcade™ 1.3 mg/m2 IV days 1 and 4 of weeks 1, 2, 4, 5, 7, 8, 10, 11, 13, and 14
  Interventions: Drug: Velcade; Drug: Rituximab

INTERVENTIONS:
Drug: Velcade — Induction: 1.3 mg/m2 IV days 1 and 4 of weeks 1, 2, 4, 5, 7, 8, 10, 11, 13 & 14.
  Maintenance: 1.3 mg/m2 IV day 1 weekly x 2 weeks beginning week 20 and continuing every 6 months until month 23.
  Other Names: Bortezomib; PS-341
Drug: Rituximab — Induction: 375 mg/m2 IV day 1 of weeks 4, 5, 7, 8, 10, 11, 13 and 14 prior to Velcade administration.
  Maintenance: 375 mg/m2 day 1 weekly x 4 weeks.
  Other Names: Rituxan

SUMMARY:
This study will determine the overall response rate and toxicity of rituximab and Velcade in combination in patients with relapsed or refractory mantle cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Rationale: Previous studies testing bortezomib and rituximab separately indicate these agents have some efficacy against mantle cell lymphoma (MCL). Bortezomib is a targeted cancer drug that blocks proteasomes. The proteasome is an enzyme complex existing in all cells that influences proteins controlling cellular processes. By blocking the proteasome, bortezomib disrupts biologic pathways such as those related to the growth and survival of cancer cells. Rituximab is a monoclonal antibody that attaches to a protein called the CD20 antigen that is found almost exclusively on the surface of B-cells with leukemia. Once rituximab attaches to the protein, the immune system activates to kill the malignant B-cells. The current study combines bortezomib and rituximab in patients with relapsed or refractory MCL.

Purpose: This study will evaluate the safety and efficacy of bortezomib and rituximab in patients with relapsed or refractory MCL. Blood, molecular, and tumor analysis will be conducted to provide researchers with information about areas such as rituximab resistance, the effects of bortezomib on cells associated with immune function, and protein alterations related to the cellular growth and death of MCL. In addition, the role of maintenance therapy and timing of administration in MCL will be assessed.

Treatment: Patients in this study will receive bortezomib and rituximab. Both drugs will be administered through intravenous infusions. There are two treatment periods in this study. The first is considered induction therapy where patients will receive bortezomib and rituximab intermittently over an eighteen week period. Lower dosages of rituximab will be given to patients at the beginning of the study to ensure no severe toxicity occurs. Those patients without disease growth after the eighteen weeks of treatments will continue with maintenance therapy. During this time period, patients will be given bortezomib and rituximab for up to one year and a half. Several tests and exams will be conducted throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell or follicular lymphoma
* Relapsed or refractory disease
* ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, 2 or 3

Exclusion Criteria:

* Pre-existing sensory or motor peripheral neuropathy
* No active or untreated CNS (Central Nervous System) lymphoma
* History of severe, life-threatening hypersensitivity or infusion reactions prior rituximab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, MD, Principal Investigator — The Ohio State University Comprehensive Medical Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Baiocchi RA, Alinari L, Lustberg ME, Lin TS, Porcu P, Li X, Johnston JS, Byrd JC, Blum KA. Phase 2 trial of rituximab and bortezomib in patients with relapsed or refractory mantle cell and follicular lymphoma. Cancer. 2011 Jun 1;117(11):2442-51. doi: 10.1002/cncr.25792. Epub 2010 Dec 14. PMID 24048792
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2005 until June 2009, 25 patients aged ≥ 18 years with historically confirmed, grade 1 or 2 mantel cell or follicular NHL according to the World Health Organization classification who relapsed or were refractory after at least 1 previous therapy.
Period: Overall Study
Arm/Group | Velcade and Rituximab
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Velcade and Rituximab
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25
Lymphoma Disease Stages [Number; unit: participants] — Ann Arbor staging system
  participants
    I(lymph node area or 1 organ outside lymph system | 2
    II(2 or more groups of lymph nodes) | 1
    Stage III(lymph node areas on both sides) | 9
    IV(outside lymph system into organ) | 13
B-symptoms [Number; unit: participants]
  Yes | 6
  No | 19
Disease Type [Number; unit: participants]
  Mantle cell lymphoma | 14
  Follicular lymphoma | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall survival in patients with relapsed or refractory mantle cell and follicular lymphoma following treatment with rituximab and Velcade™.
Time Frame: Every 3 months
Measure: Number; unit: percentage of patients
Arm/Group | Velcade and Rituximab
Number analyzed (Participants) | 25
percentage of patients
  All patients | 40
  Patients with follicular lymphoma | 55
  Patients with MCL | 29

2. Primary Outcome: Assess the Toxicity of Combination Rituximab and Velcade™ in Patients With Previously Treated Mantle Cell and Follicular Lymphoma.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for adverse event reporting.
Time Frame: Day 1 of each cycle
Population: grade 3 neurotoxicity which consisted of constipation/ileus, sensory or motor neuropathy, or orthostatic hypotension
Measure: Number; unit: patients
Arm/Group | Velcade and Rituximab
Number analyzed (Participants) | 25
patients | 13

3. Secondary Outcome: Progression-free Survival(PFS)
Description: To correlate serial plasma rituximab levels with response and progression-free survival.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Velcade and Rituximab
Number analyzed (Participants) | 25
percentage of patients
  All patients | 24 [10 to 53]
  Responding patients | 60 [20 to 85]

4. Secondary Outcome: Correlative Studies
Time Frame: During induction (weeks 1-15); PK every 2 months during maintenance.
Population: Data not collected and analyzed
Groups:
- Velcade and Rituximab: Rituximab 375 mg/m2 IV day 1 of weeks 4, 5, 7, 8, 10, 11, 13, and 14 prior to Velcade™ administration.
  Velcade™ 1.3 mg/m2 IV days 1 and 4 of weeks 1, 2, 4, 5, 7, 8, 10, 11, 13, and 14
  Velcade: Induction: 1.3 mg/m2 IV days 1 and 4 of weeks 1, 2, 4, 5, 7, 8, 10, 11, 13 & 14.
  Maintenance: 1.3 mg/m2 IV day 1 weekly x 2 weeks beginning week 20 and continuing every 6 months until month 23.
  Rituximab: Induction: 375 mg/m2 IV day 1 of weeks 4, 5, 7, 8, 10, 11, 13 and 14 prior to Velcade administration.
  Maintenance: 375 mg/m2 day 1 weekly x 4 weeks.
Arm/Group | Velcade and Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Velcade and Rituximab
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 25/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade and Rituximab (N=25)
Neutropenia (General disorders) | 3 (3) — Grade 3
Anemia (Blood and lymphatic system disorders) | 2 (2) — Grade 3
Thrombocytopenia (Injury, poisoning and procedural complications) | 2 (2) — Grade 3
Anorexia (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3
Sensory Neuropathy (Musculoskeletal and connective tissue disorders) | 9 (9) — Grade 3
Motor Neuropathy (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Autonomic neuropathy (Nervous system disorders) | 3 (3) — Grade 3 orthostatic hypotension
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Fatigue (General disorders) | 8 (8) — Grade 3
Myositis/Creatinine kinase elevation (Investigations) | 1 (1) — Grade 3
nausea/vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3
Constipation/ileus (Gastrointestinal disorders) | 3 (3) — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No